CLINICAL TRIAL: NCT06584201
Title: Effects of Erector Spina Plane Block and Paravertebral Block on Early Postoperative Pulmonary Function Test Parameters in Patients Undergoing Video-assisted Thoracoscopic Surgery
Brief Title: Effects of Erector Spina Plane Block and Paravertebral Block on Early Postoperative Pulmonary Function Test Parameters
Status: Recruiting | Type: Observational
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Principal Investigator, Ozal Adiyeke, director, Başakşehir Çam & Sakura City Hospital
Other Study IDs: E-96317027-514.10-222446069
Record Dates: First submitted 2024-08-09; First posted 2024-09-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Respiratory Function Loss; Pain, Postoperative; Opioid Use
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ESP Group: Patients in this group will receive the Erector Spinae Plane Block (ESP) as a method of postoperative pain management.
  Interventions: Procedure: Erector Spinae Plane Block (ESP)
- Paravertebral Group: Patients in this group will receive the Paravertebral Block (PVB) for postoperative pain relief.
  Interventions: Procedure: Paravertebral Block (PVB)

INTERVENTIONS:
Procedure: Erector Spinae Plane Block (ESP) — The ESP block will be administered before the VATS procedure, aiming to manage postoperative pain and minimize the impact on early lung function test (SFT) parameters. The block will be performed using standard techniques under ultrasound guidance to ensure accurate placement.
  Groups: ESP Group
Procedure: Paravertebral Block (PVB) — The PVB will be administered prior to the VATS procedure, with the objective of managing postoperative pain and assessing its impact on early postoperative lung function (SFT) parameters. This block will also be performed using standard techniques and ultrasound guidance for precision.
  Groups: Paravertebral Group

SUMMARY:
The pain experienced by participants after minimally invasive chest surgery (VATS) can make it difficult for them to take deep breaths, which can lead to problems with lung function. This can cause serious problems such as lung collapse, low oxygen levels, and infections, making recovery longer and more difficult. Managing pain well after surgery is important to prevent these problems and speed up recovery. In this study, we aimed to compare two pain relief methods, Erector Spinae Plane Block (ESP) and Paravertebral Block (PVB), in participants who underwent VATS. We will look at which method causes the smallest change in lung function before and after surgery.

DETAILED DESCRIPTION:
Video-assisted Thoracoscopic surgery (VATS) is a minimally invasive surgical method used in the diagnosis and treatment of diseases in the chest area. Thoracoscopic surgery has many advantages, such as being less invasive, less risk of complications, shorter hospital stay, and better cosmetic results. However, these participants may experience severe pain in the postoperative period, although not as much as in surgeries performed with open surgical methods, that is, thoracotomy. This pain, which occurs in the postoperative period in VATS methods, which is one of the minimally invasive methods, may prevent the participants from taking deep breaths, as well as cause deterioration of respiratory functions, serious pulmonary complications such as atelectasis, hypoxia and infection, and prolonged postoperative patient stay. As the development of morbidity and mortality. Delay or deterioration in postoperative respiratory functions is one of the most troublesome complications of thoracic surgery. It was reported that acute pain in the postoperative period should be effectively controlled with effective analgesia methods in order to prevent postoperative pulmonary complications and accelerate the patient's well-being. Controlling pain with postoperative analgesia allows participants to breathe more deeply, perform breathing exercises more effectively, and therefore improves and helps preserve respiratory functions. Although thoracic epidural analgesia is the gold standard method in thoracic surgery, intravenous analgesic techniques and thoracic trunk nerve blocks are increasingly recommended for postoperative analgesia in less invasive VATS operations. Thoracic trunk blocks have effects on hemodynamics, respiratory functions, and consciousness; It has important advantages such as having fewer side effects than systemic analgesic techniques and being less invasive than thoracic epidural analgesia. Body blocks are recommended as a first-line analgesia program, especially in thoracic surgery, as they shorten postoperative recovery time, reduce the risk of pneumonia and provide early postoperative mobilization. The ease of application of the erector spinae plane block (ESP), its low risk of complications, and its ability to provide effective analgesia, especially in minimally invasive surgeries, have increased its use. Paravertebral block (PVB), one of the other blocks, is frequently used because it is more reliable and provides effective analgesia compared to thoracic epidural analgesia and conventional analgesia methods. Thoracic trunk plane blocks can significantly reduce intravenous opioid use and prevent side effects related to opioid use with the effective analgesia they provide in the early postoperative period, increase participants' comfort and painlessness, and accelerate recovery while preventing deterioration in respiratory function parameters. during rest and mobilization. Because; It is thought that by applying erector spinae plane block (ESP) or paravertebral block (PVB), postoperative pain scores and opioid consumption will decrease significantly and respiratory functions will return earlier. In this study, we aimed to evaluate the effects of ESP or PVB on respiratory functions in the early postoperative period in patients undergoing VATS, and in which block there would be less percentage change between preoperative and postoperative respiratory function test (PFT) parameters.

Pain is a symptom known to be subjective and will be queried with a standardized scale, the visual pain score scale (VAS), to minimize differences between participants. Postoperative rest and movement pain scores (VAS; 0, 1, 2, 4, 6, 12, 24 and pre-discharge scores), postoperative 6th hour, 24th hour and predischarge pulmonary function test (PFT) parameters, total Analgesic consumption will be recorded at 0, 1, 2, 4, 6, 12, 24 hours and before discharge.

Forced Vital Capacity (FVC), Forced Expiratory Volume in 1 Second (FEV1), FEV1/FVC, Peak Expiratory Flow (PEF) values will be recorded as Respiratory Function Test parameters.

The total narcotic analgesic needs of the participants who received the block will be recorded with the PCA device placed intravenously postoperatively and their total Morphine consumption will be recorded.

Participants' satisfaction after the procedure will be questioned with a Likert score before discharge.

Side effects such as nausea and vomiting that may occur in participants will be questioned with the simplified post-operative nausea and vomiting impact scale.

Participants' demographic characteristics, comorbidities, operation times and complications will be recorded and statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Both genders
* Being between the ages of 18 and 65
* ASA(American Society of Anesthesiologists) I-II-III
* Body mass index between 19 and 30kg/m2
* Providing voluntary participation
* Must be fully oriented and able to cooperate

Exclusion Criteria:

* ASA(American Society of Anesthesiologists) IV-V
* Patients who refuse to participate in the study
* Patients under 18 years of age
* Patients over 65 years of age
* Presence of active infection in the area to be treated
* Chronic pain and constant analgesic use
* Patients with coagulation disorders
* Patients who cannot cooperate with postoperative pain follow-ups
* Cases taken urgently
* Patients with severe renal failure (creatinine>2mg/dl)
* Severe impairment of heart function (New York Heart Association Functional Classification III-IV)
* Patients with known allergies to bupivacaine and other amide local anesthetic substances.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants aged 18-65 who will undergo video-assisted thorascopic surgery
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Effectiveness on respiratory functions | Respiratory function tests will be performed 24 hours before surgery and at 0, 6, and 24 hours postoperatively, as well as before discharge. The average length of stay is 2 days, and for extended stays, the 48-hour data will be used as a baseline.
  All adult participants undergoing video-assisted thoracoscopic surgery (VATS) will have a preoperative pulmonary function test (PFT) conducted by an anesthetist using a portable device within the Thoracic Surgery service. The tests will be evaluated using a color-coded compliance chart: Red (Non-compliant), Yellow (Moderately compliant), Green (Compliant). The test will be repeated until compliance is achieved, with Yellow and Green results recorded. Postoperatively, PFTs will be repeated at 0, 6, 24 hours, and before discharge. The specific pulmonary function tests assessed include Forced Vital Capacity (FVC), Forced Expiratory Volume in 1 second (FEV1), Peak Expiratory Flow (PEF), Forced Expiratory Flow at 25-75% (FEF25-75), and the FEV1/FVC ratio. Each test will be reported as separate outcome measures. Respiratory function tests will be conducted 24 hours before surgery and then postoperatively at the specified intervals.

SECONDARY OUTCOMES:
Effect on total narcotic analgesic consumption | Total dose administered at the end of 24 hours of the intravenous PCA device inserted simultaneously after surgery
  After the surgery, participants will receive intravenous patient-controlled analgesia (PCA) and infusion will begin simultaneously with the end of the operation. "Morphine" was preferred as the treatment method to be used in the PCA method. In PCA preparation, 30 mg morphine is added to 100 cc of physiological saline. As the PCA protocol, 3 mg loading dose, 1 cc/hour (0.3 mg/hour) basal infusion dose, 3 cc (1 mg) bolus dose, 10-minute lockout period (maximum 2 bolus doses in 1 hour) were set. The total number of bolus doses administered by the participants on the PCA device at the end of 24 hours will be recorded and evaluated as the amount of additional opioid needed.

OTHER OUTCOMES:
Effectiveness on pain scores | 0, 1, 4, 6, 12 and 24 hours after surgery
  Postoperative pain assessment is made using visual pain scoring. Participants are asked about their resting pain 0, 1, 4, 6, 12 and 24 hours after applying a postoperative peripheral nerve block. With this method, participants rate their pain with a precise numerical value from 0 to 10. While zero(0) represents "no pain"; Ten (10) represents the opposite end of the pain continuum (e.g., "The most intense pain imaginable," "As intense pain as possible," "unbearable pain").

CONTACTS AND LOCATIONS:
Locations (1):
- Basaksehir Çam Ve Sakura City Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Result] Matyal R, Montealegre-Gallegos M, Shnider M, Owais K, Sakamuri S, Shakil O, Shah V, Pawlowski J, Gangadharan S, Hess P. Preemptive ultrasound-guided paravertebral block and immediate postoperative lung function. Gen Thorac Cardiovasc Surg. 2015 Jan;63(1):43-8. doi: 10.1007/s11748-014-0442-6. Epub 2014 Jul 1. PMID 24980146
- [Result] Detterbeck FC. Efficacy of methods of intercostal nerve blockade for pain relief after thoracotomy. Ann Thorac Surg. 2005 Oct;80(4):1550-9. doi: 10.1016/j.athoracsur.2004.11.051. PMID 16181921
- [Result] Gao W, Yang XL, Hu JC, Gu H, Wu XN, Hu SS, Wang S, Chai XQ, Wang D. Continuous Serratus Anterior Plane Block Improved Early Pulmonary Function After Lung Cancer Surgical Procedure. Ann Thorac Surg. 2022 Feb;113(2):436-443. doi: 10.1016/j.athoracsur.2021.02.032. Epub 2021 Mar 2. PMID 33667460
- [Result] Zengin M, Baldemir R, Ulger G, Sazak H, Alagoz A. Postoperative Analgesic Efficacy of Thoracic Paravertebral Block and Erector Spinae Plane Block Combination in Video-Assisted Thoracic Surgery. Cureus. 2021 Jun 12;13(6):e15614. doi: 10.7759/cureus.15614. eCollection 2021 Jun. PMID 34277232